CLINICAL TRIAL: NCT06952647
Title: Evaluation of Inflammatory Hematological Markers in Idiopathic Carpal Tunnel Syndrome
Brief Title: Hematological Markers in Idiopathic Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nadide Koca, Principal Investigator, Ankara Training and Research Hospital
Other Study IDs: AnkaraTRH-FTR-NK-04
Record Dates: First submitted 2025-04-19; First posted 2025-05-01 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Carpal Tunnel Syndrome (CTS); Biomarkers / Blood
Keywords: Carpal Tunnel Syndrome (CTS); Vitamin b12; Biomarkers / blood
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case-Idiopathic Carpal Tunnel Syndrome Patient Group: Patients diagnosed with idiopathic Carpal Tunnel Syndrome, confirmed by electrodiagnostic testing, with no identifiable secondary causes. Evaluated for inflammatory hematological markers and vitamin B12 levels.
- Control- Healthy Control Group (Electrodiagnostically Screened): Age- and sex-matched asymptomatic individuals without Carpal Tunnel Syndrome, confirmed through electrodiagnostic testing. Used as controls for comparison of inflammatory markers and vitamin B12 levels.

SUMMARY:
Carpal Tunnel Syndrome (CTS) cases are still classified as idiopathic. The rationale of this research is to investigate the role of chronic inflammation and vitamin B12 deficiency in the onset and severity of idiopathic CTS. This case-control study aims to evaluate inflammatory hematological markers and vitamin B12 levels in patients with idiopathic CTS compared to healthy controls, and to analyze their correlation with clinical and electrophysiological severity of the disease

DETAILED DESCRIPTION:
The carpal tunnel, located on the palmar side of the wrist, is bounded medially by the pisiform and hook of hamate, and laterally by the tuberosities of scaphoid and trapezium. The thick connective tissue (flexor retinaculum) covers these four bony prominences, forming a tunnel for the extrinsic flexor tendons of the fingers (flexor digitorum profundus, flexor digitorum superficialis, and flexor pollicis longus), keeping them in place during wrist flexion. The median nerve is the major peripheral nerve of the upper extremity. It originates from the lateral and medial cords of the brachial plexus. It progresses along the arm to the forearm, following a path through the carpal tunnel toward the wrist; here, it branches to provide motor support to the thenar muscle group and sensory innervation to the palmar surface. It innervates the thumb, index finger, middle finger, and half of the ring finger. Carpal Tunnel Syndrome (CTS) occurs when the tunnel narrows or the extrinsic flexor tendons or tendon sheaths swell. It is most commonly seen in the 3rd-5th decades and is three times more common in women than men. The narrowing in the carpal tunnel affects the median nerve, causing sensory disturbance symptoms in the innervated fingers. Symptoms can progress to thenar muscle weakness, leading to weakened grip strength.

Although the pathophysiology of CTS is multifactorial, it can be simplified as compression of the median nerve at the carpal tunnel level. The two most common compression sites are under the flexor retinaculum at the tunnel exit and the hook of hamate. Compression results from increased compartmental pressure in the carpal tunnel and decreased volume. The most common mechanism is hypertrophy of the synovial tissue surrounding the extrinsic flexor tendons of the hand. This hypertrophy may develop due to overuse, wrist trauma, or an underlying inflammatory process such as arthritis. Systemic diseases such as obesity, diabetes mellitus (DM), chronic kidney disease, rheumatoid arthritis, hypothyroidism, congestive heart failure, and pregnancy are also risk factors for CTS.

High body mass index (BMI) is a significant risk factor in developing CTS. A positive correlation between BMI and CTS severity has been reported. CTS is more common in patients with metabolic syndrome, which is characterized by abdominal obesity, atherogenic dyslipidemia, high blood pressure, insulin resistance or glucose intolerance, and is a prothrombotic and proinflammatory endocrinopathy. CTS severity is also higher in these patients.

Environmental workplace factors may promote the development of carpal tunnel syndrome. There is evidence that high levels of repetitive wrist movement increase the risk of carpal tunnel syndrome. There are dramatic changes in fluid pressure in the carpal tunnel according to wrist position; extension increases pressure 10-fold, and wrist flexion increases it 8-fold. Additionally, certain workplace psychosocial factors such as high psychological job demands, high job strain, low level of autonomy over one's work, and absence of interpersonal relationships providing social support are reported to be associated with carpal tunnel syndrome.

Despite various risk factors mentioned above, most CTS cases are still idiopathic cases where the cause cannot be determined. Therefore, comprehensive studies on pathophysiology and etiology continue. In CTS, which can lead to serious disability, a single factor often cannot explain the etiology. Therefore, many risk factors remain unidentified.

In idiopathic CTS, a pathophysiology that triggers each other in the form of ischemia, oxidative stress, low-grade chronic inflammation, and fibrosis, further narrowing the tunnel is emphasized.

In recent years, based on the knowledge that chronic inflammation creates an imbalance in peripheral blood neutrophil, lymphocyte, platelet, and monocyte counts, certain hematological indices have been developed by comparing these blood cells to each other. Commonly used ones are neutrophil/lymphocyte ratio (NLR), platelet/lymphocyte ratio (PLR), monocyte/lymphocyte ratio (MLR), systemic immune inflammation index (SII) calculated by platelet count X neutrophil count/lymphocyte count formula, and systemic immune response index (SIRI) calculated by neutrophil count X monocyte count/lymphocyte count formula. These indices are reported as simple and useful markers reflecting chronic inflammation in many diseases. In a study conducted with routine hemogram parameters in patients with idiopathic CTS, an increased neutrophil/lymphocyte ratio (NLR) was reported to correlate with CTS severity, and in another study, elevated CRP was reported to correlate with CTS severity, emphasizing systemic inflammation in the etiology of idiopathic CTS.

CTS is the most common cause of acroparesthesia. However, apart from systemic diseases, vitamin B12 deficiency is also an important cause. In a study comparing risk factors between moderate CTS and severe CTS patient groups, no difference was found in terms of age, gender, occupational risk factors, and systemic diseases such as DM, hypothyroidism, rheumatoid arthritis, cardiovascular disease, and renal failure. On the other hand, the same study reports that high BMI and vitamin B12 deficiency were significantly higher in the severe CTS group than in the moderate CTS group.

Despite numerous evidences reached through studies, most CTS cases are still classified as idiopathic. This research aims to investigate the role of chronic inflammation and vitamin B12 deficiency in the onset and severity of idiopathic CTS.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* Having undergone Electromyography (EMG) testing for Carpal Tunnel Syndrome (CTS)-like symptoms
* Recent complete blood count, C-Reactive Protein (CRP), and vitamin B12 tests available

Exclusion Criteria:

* Age below 18 or above 65 years
* Pregnancy
* History of wrist trauma or surgical operation
* Diabetes mellitus
* Chronic kidney disease
* Gout
* Rheumatoid arthritis
* Connective tissue disease
* Thyroid disorders
* Acromegaly
* Polyneuropathy
* Thoracic outlet syndrome
* Brachial plexopathy
* Cervical disc herniation
* Presence of cardiac pacemaker
* Steroid use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Electromyography (EMG) laboratory/clinic with suspected Carpal Tunnel Syndrome (CTS) who underwent electrodiagnostic testing
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of Systemic Inflammation Response Index (SIRI) as an Inflammatory Marker | up to 4 weeks
  The systemic inflammation response index (SIRI) is calculated as neutrophil count × monocyte count / lymphocyte count. It reflects the combined effect of neutrophil and monocyte-driven innate immunity versus lymphocyte-mediated adaptive immunity. SIRI has been proposed as a robust marker of inflammation in several chronic diseases.
  In the current study, SIRI was evaluated in individuals with and without Carpal Tunnel Syndrome (CTS) to investigate its potential as an indicator of inflammatory burden.

SECONDARY OUTCOMES:
Comparison of vitamin B12 | up to 4 weeks
  Comparison of vitamin B12 levels between case and control groups
Evaluation of Electromyography severity | up to 4 weeks
  EMG (Electromyography) intensity/amplitude is an important parameter used in the electrical measurement of muscle activity. Electromyography (EMG) severity;
  * Mild: Minimal abnormalities with slight spontaneous activity and minor changes in motor unit potentials
  * Moderate: Significant spontaneous activity with noticeable changes in recruitment patterns
  * Severe: Extensive spontaneous activity (fibrillations, positive sharp waves), significant reduction or increase in motor unit potentials, and severe recruitment abnormalities
- Comparison of C-Reactive Protein levels (CRP) | up to 4 weeks
  - Comparison of C-Reactive Protein levels (CRP) levels between case and control groups. CRP is an acute phase protein used as an inflammatory marker. CRP's half-life is approximately 19 hours, making it a responsive marker that can indicate both the onset of inflammation and the response to treatment relatively quickly.
Evaluation of Platelet/Lymphocyte Ratio (PLR) as an Inflammatory Marker | up to 4 weeks
  Platelet/lymphocyte ratio (PLR) is another hematological marker that reflects systemic inflammation. During inflammatory responses, platelet counts often increase while lymphocyte counts decrease, resulting in an elevated PLR. Platelets play an active role in inflammation by releasing inflammatory mediators and interacting with leukocytes. PLR, calculated from routine blood tests, has been increasingly used in the assessment of inflammatory conditions.
  In this study, PLR values were compared between patients with Carpal Tunnel Syndrome (CTS) and healthy controls to evaluate its association with inflammation in CTS.
Evaluation of Monocyte/Lymphocyte Ratio (MLR) as an Inflammatory Marker | up to 4 weeks
  Monocyte/lymphocyte ratio (MLR) is a peripheral blood marker used to assess systemic inflammatory status. Monocytes contribute to chronic inflammation and tissue remodeling, while lymphocytes are typically reduced in inflammatory states. An increased MLR may reflect an enhanced inflammatory response. Like other ratios, MLR can be easily derived from complete blood count parameters.
  In this study, MLR was analyzed in patients with and without Carpal Tunnel Syndrome (CTS) to explore its relevance as a potential inflammatory biomarker.
Evaluation of Neutrophil/Lymphocyte Ratio (NLR) as an Inflammatory Marker | up to 4 weeks
  In inflammatory diseases, the immune response often leads to an increase in circulating neutrophils and a decrease in lymphocytes, resulting in an elevated neutrophil/lymphocyte ratio (NLR). This parameter has recently gained attention as a simple, cost-effective, and readily available marker of systemic inflammation. NLR is derived from routine complete blood count tests and reflects the balance between innate (neutrophils) and adaptive (lymphocytes) immune responses.
  In the present study, NLR was compared between patients with Carpal Tunnel Syndrome (CTS) and healthy controls to investigate its potential role as a marker of inflammation in CTS.
Evaluation of Systemic Immune-inflammation Index (SII) as an Inflammatory Marker | up to 4 weeks
  The systemic immune-inflammation index (SII) is a composite marker calculated using the formula: platelet count × neutrophil count / lymphocyte count. It simultaneously incorporates three types of immune cells and is considered a more comprehensive indicator of the systemic inflammatory status. Elevated SII levels have been associated with various inflammatory and immune-mediated conditions.
  In this study, SII values were compared between CTS patients and healthy controls to assess its potential utility in identifying inflammatory activity in CTS.

CONTACTS AND LOCATIONS:
Overall Officials: Nadide Koca, M.D., Principal Investigator — University of Health Sciences, Ankara Training and Research Hospital, TURKEY
Locations (1):
- Department of Physical Therapy and Rehabilitation, University of Health Sciences, Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional policies regarding patient privacy and data protection regulations

REFERENCES:
- [Background] Tonga F, Bahadir S. The Factors Associated with Carpal Tunnel Syndrome Severity. Turk Neurosurg. 2022;32(3):392-397. doi: 10.5137/1019-5149.JTN.34519-21.2. PMID 34859834
- [Background] Zvonickova K, Rhee A, Sandy-Hindmarch O, Furniss D, Wiberg A, Schmid AB. Systemic low-grade C-reactive protein is associated with proximal symptom spread in carpal tunnel syndrome. Pain Rep. 2024 Apr 10;9(3):e1156. doi: 10.1097/PR9.0000000000001156. eCollection 2024 Jun. PMID 38606315
- [Background] Gunes M, Buyukgol H. Correlation of neutrophil/lymphocyte and platelet/lymphocyte ratios with the severity of idiopathic carpal tunnel syndrome. Muscle Nerve. 2020 Mar;61(3):369-374. doi: 10.1002/mus.26791. Epub 2020 Jan 9. PMID 31875987
- [Background] Wang RH, Wen WX, Jiang ZP, Du ZP, Ma ZH, Lu AL, Li HP, Yuan F, Wu SB, Guo JW, Cai YF, Huang Y, Wang LX, Lu HJ. The clinical value of neutrophil-to-lymphocyte ratio (NLR), systemic immune-inflammation index (SII), platelet-to-lymphocyte ratio (PLR) and systemic inflammation response index (SIRI) for predicting the occurrence and severity of pneumonia in patients with intracerebral hemorrhage. Front Immunol. 2023 Feb 13;14:1115031. doi: 10.3389/fimmu.2023.1115031. eCollection 2023. PMID 36860868
- [Background] Malakootian M, Soveizi M, Gholipour A, Oveisee M. Pathophysiology, Diagnosis, Treatment, and Genetics of Carpal Tunnel Syndrome: A Review. Cell Mol Neurobiol. 2023 Jul;43(5):1817-1831. doi: 10.1007/s10571-022-01297-2. Epub 2022 Oct 10. PMID 36217059
- [Background] Padua L, Cuccagna C, Giovannini S, Coraci D, Pelosi L, Loreti C, Bernabei R, Hobson-Webb LD. Carpal tunnel syndrome: updated evidence and new questions. Lancet Neurol. 2023 Mar;22(3):255-267. doi: 10.1016/S1474-4422(22)00432-X. Epub 2022 Dec 13. PMID 36525982
- [Background] Werner RA, Andary M. Carpal tunnel syndrome: pathophysiology and clinical neurophysiology. Clin Neurophysiol. 2002 Sep;113(9):1373-81. doi: 10.1016/s1388-2457(02)00169-4. PMID 12169318
- [Background] Otelea MR, Nartea R, Popescu FG, Covaleov A, Mitoiu BI, Nica AS. The Pathological Links between Adiposity and the Carpal Tunnel Syndrome. Curr Issues Mol Biol. 2022 Jun 8;44(6):2646-2663. doi: 10.3390/cimb44060181. PMID 35735622
- [Background] Joshi A, Patel K, Mohamed A, Oak S, Zhang MH, Hsiung H, Zhang A, Patel UK. Carpal Tunnel Syndrome: Pathophysiology and Comprehensive Guidelines for Clinical Evaluation and Treatment. Cureus. 2022 Jul 20;14(7):e27053. doi: 10.7759/cureus.27053. eCollection 2022 Jul. PMID 36000134
- [Background] Newington L, Harris EC, Walker-Bone K. Carpal tunnel syndrome and work. Best Pract Res Clin Rheumatol. 2015 Jun;29(3):440-53. doi: 10.1016/j.berh.2015.04.026. Epub 2015 May 27. PMID 26612240